CLINICAL TRIAL: NCT05347615
Title: The Implantation Of Monofocal And Premium IOL Models - A Registry Study At The Kepler University Hospital
Brief Title: Achieving Hybrid Monovision By Paring Monofocal And EDOF Lens Technology
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Matthias Bolz, Head of Ophthalmology, Johannes Kepler University of Linz
Other Study IDs: KUK-Ophthalmology-006
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EDOF: Eye after EDOF lens Implantation
  Interventions: Procedure: IOL Implantation:EDOF lens
- Monofocal: Eye after Monofocal lens Implantation
  Interventions: Procedure: IOL Implantation: Monofocal lens

INTERVENTIONS:
Procedure: IOL Implantation:EDOF lens — A EDOF lens is implanted in the dominant eye
  Groups: EDOF
Procedure: IOL Implantation: Monofocal lens — A monofocal lens is implanted in the non dominant eye.
  Groups: Monofocal

SUMMARY:
Modern day cataract surgery isn't just a rehabilitative procedure anymore but rather aims at improving a patient's quality of life by reducing the need for spectacles in everyday life to a minimum. One way of achieving this goal is by using different lens technologies, such as a monofocal lens paired a lens with EDOF technology, as EDOF lenses provide an enhanced depth of focus by creating a single elongated focal point. As this "mix-and-match" is well established, the aim of this study is to compare the monofocal lens cohort to the EDOF lens cohort and evaluate visual acuity and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 21-99 years
* signed consent form
* senile cataract LOCS III grading
* Cataract surgery with monofocal or premium lens implantation

Exclusion Criteria:

* missing signed consent form
* macular pathologies
* corneal pathologies
* irregular astigmatism
* pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients with senile cataract undergoing surgery
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
uncorrected distance visual acuity | 24 months
  Percentage of patients with uncorrected distance visual acuity of logMAR >0.1
uncorrected intermediate distance visual acuity | 24 months
  Percentage of patients with uncorrected intermediate distance visual acuity of logMAR >0.2
uncorrected near visual acuity | 24 months
  Percentage of patients with uncorrected near visual acuity of logMAR >0.2

SECONDARY OUTCOMES:
Dysphotopsia | 24 months
  Quality of Vision questionnaire
PRISQ-Questionnaire | 24 months
  questionnaire rating spectacle independency
Patient Satisfaction | 24 months
  Catquest 9-SF-Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Kepler University, Linz, Austria

IPD SHARING:
Plan to Share IPD: No